CLINICAL TRIAL: NCT05828862
Title: Investigating the Effect of Hypotension Prediction Index Guidance on Intraoperative Hypotension and the Relationships Between the Metabolomic Profile and Postoperative Ileus in Patients Undergoing Major Upper Abdominal Surgery: a Randomized Controlled Trial
Brief Title: Intraoperative Hypotension and Metabolomics in Major Upper Gastrointestinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202301110DIND
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: the Intraoperative Hypotension

STUDY DESIGN:
Intervention Model Description: patients undergoing Hypotension Prediction Index
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypotension prediction index guided (Experimental): patients with hypotension prediction index guidance
  Interventions: Procedure: hypotension prediction index guidance

INTERVENTIONS:
Procedure: hypotension prediction index guidance — using hypotension prediction index guidance to prevent intraoperative hypotension

SUMMARY:
We will investigate the effect of hypotension prediction index guidance on intraoperative hypotension and metabolomics in patients undergoing major upper gastrointestinal surgery

DETAILED DESCRIPTION:
Intraoperative hypotension (IOH) has been shown to increase the risk of postoperative morbidity and mortality. The Hypotension prediction index (HPI) guidance is an algorithm that can predict impending hypotension, defined as mean arterial pressure below 65mmHg. Patients undergoing major upper abdominal surgery are at high risk of IOH occurrence, because the surgical procedures involve organ removal like intestinal resection and vessel or organ anastomoses or reconstruction, often associated with high blood loss. However, the effectivity of applying HPI for reducing the duration and severity of IOH and postoperative morbidity and mortality in short term within 30 days after surgery and long term within 1 year remains inconclusive.

Postoperative ileus (POI) generally defines absence of flatus within 72 hours after surgery. POI is known as the most important factor to slow patient recovery, increase postoperative morbidity and prolong the hospital stay following major upper abdominal surgery. Metabolomics can investigate the small molecule changes in response to certain stimulus, such as different environments. Metabolomics involves the comprehensive analysis of metabolites. In recent years, metabolomics has several applications in the early diagnosis and prevention of health and disease. However, the association between the POI occurrence and the metabolites in the presence and absence HPI guidance have not yet been investigated.

The proposed strategy and specific objectives of this 2 years project using a randomized controlled trial are as the follows:

1. To clarify the relationship of POI occurrence to presence and absence of HPI guidance
2. To Explore differences in metabolites in presence or absence of HPI guidance.
3. Explore the potential metabolites associated with POI in different intraoperative environment in using HPI and no HPI guidance.

ELIGIBILITY:
Inclusion Criteria:

* elective upper gastrointestinal surgery

Exclusion Criteria:

* no laparoscopic surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-04-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
time weighted average mean arterial pressure less than 65 mmHg | surgery
  the severity and duration of hypotension during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
due to ethical issue